CLINICAL TRIAL: NCT05987124
Title: A Phase II Intrapatient Open-Label Dose Escalation Trial of Defibrotide in Hematopoietic Cell Transplantation (HCT) Recipients With Sinusoidal Obstructive Syndrome (SOS) Post-HCT Associated With Either Renal and/or Pulmonary Dysfunction With Either Refractory or Progressive Disease Following Defibrotide Therapy
Brief Title: Defibrotide Dose-escalation for SOS Post-HSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 600
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Sinusoidal Obstruction Syndrome; Veno-occlusive Disease
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Defibrotide (Experimental): 7.1.1 HCT recipients with SOS/VOD and renal and/or pulmonary dysfunction with either PR after 21 days of standard doses of defibrotide (25mg/kg/day) or SD, after 14 days of standard doses of defibrotide (25mg/kg/day) progressive disease after 7 days on defibrotide (25mg/kg/day) will undergo intra-patient dose escalation every 4 days until a complete response is obtained up until the highest dose level of 100mg/kg/day at which point an endpoint of CR, PR or SD will be sought (see 7.2 for definition of response) (Maximum of 4 dose levels) (7.1.2):
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — HCT recipients with SOS/VOD and renal and/or pulmonary dysfunction with either PR after 21 days of standard doses of defibrotide (25mg/kg/day) or SD, after 14 days of standard doses of defibrotide (25mg/kg/day) progressive disease after 7 days on defibrotide (25mg/kg/day) will undergo intra-patient dose escalation every 4 days until a complete response is obtained up until the highest dose level of 100mg/kg/day at which point an endpoint of CR, PR or SD will be sought(Maximum of 4 dose levels). Defibrotide will be administered in D5W or 0.9% NaCl via IV infusion over 2 hours q6 hours.
  Other Names: Defitelio

SUMMARY:
This research study is being done to determine the safety and tolerability of increasing doses of defibrotide within a single patient with sinusoidal obstructive syndrome (SOS)/veno-occlusive disease (VOD) after hematopoietic cell transplantation (HCT) associated with either kidney and/or lung impairment that has not obtained a complete response (CR) or progressed in severity with standard doses of defibrotide.

ELIGIBILITY:
Inclusion Criteria:

* HCT recipients (Auto or Allograft)
* SOS/VOD as defined by Cairo/Cooke Diagnostic criteria (1) (Table 3) with either renal and/or pulmonary dysfunction as defined by Cairo/Cooke Grading criteria (1) (Appendix I).
* Unresponsive to standard defibrotide therapy as defined by at least one of the following:
* Patients with SOS/VOD failing to obtain a complete response (CR) defined by Grade I or less by Cairo/Cooke Grading criteria (1) (Appendix I). This would therefore include patients with stable disease after at least 14 days of defibrotide or partial response after at least 21 days of defibrotide (25mg/kg/day).
* Progressive disease defined by progression of at least one grade or more from diagnostic grade as defined by Cairo/Cooke Grading criteria (1) (Appendix I) following at least 7 days of defibrotide (25mg/kg/day).
* Age 1 month - 75 years

Exclusion Criteria:

* Patients who did not receive HCT.
* Concomitant systemic anticoagulation (excluding central venous line management, fibrinolytic instillation for central venous line occlusion, management of intermittent dialysis or ultrafiltration of CVVH).
* Active bleeding and/or hemorrhage of at least grade 2 and above.
* History of development of Grade III/IV anaphylaxis probably or directly secondary to defibrotide.
* Female patients who are pregnant or breast feeding.

Ages: 1 Month to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of grade 3 or 4 adverse events related to defibrotide | 100 days
  grade 3 and 4 adverse events possible or probably related to defibrotide will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States